CLINICAL TRIAL: NCT06203756
Title: Improved Patient Outcomes With Robotic-Assisted Total Knee Arthroplasty
Brief Title: Patient Outcomes With Robotic-Assisted Total Knee Arthroplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSP-2017-01
Record Dates: First submitted 2023-12-11; First posted 2024-01-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Arthroplasties, Knee Replacement; Revision Arthroplasty
Keywords: Robotic-Assisted Total Knee Arthroplasty; Knee Replacement; Knee outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Revision Total Knee Arthroplasty (Other): Sensor-assisted robotic surgery cohort with a tibia first workflow. Revision Total Knee Arthroplasty components.
  Interventions: Device: Omnibotics Robotic-assisted Total Knee Arthroplasty with Apex Revision
- Primary Total Knee Arthroplasty (Other): Sensor-assisted robotic surgery cohort with a tibia first workflow. Primary Total Knee Arthroplasty
  Interventions: Device: Omnibotics Robotic-assisted Total Knee Arthroplasty with Apex UC; Device: Omnibotics Robotic-assisted Total Knee Arthroplasty with Apex PS

INTERVENTIONS:
Device: Omnibotics Robotic-assisted Total Knee Arthroplasty with Apex UC — Robotic-assisted total knee arthroplasty in femur and tibial first workflows using the BalanceBot to characterize soft tissue balance, and the Apex UltraCongruent (UC) knee implant type
  Other Names: BalanceBot, Apex Knee System, Active Spacer
  Arms: Primary Total Knee Arthroplasty
Device: Omnibotics Robotic-assisted Total Knee Arthroplasty with Apex PS — Robotic-assisted total knee arthroplasty with a tibial first workflow using the BalanceBot to characterize soft tissue balance, and the Apex PosteriorStabilized (PS) knee implant type
  Arms: Primary Total Knee Arthroplasty
Device: Omnibotics Robotic-assisted Total Knee Arthroplasty with Apex Revision — Robotic-assisted total knee arthroplasty with a tibial first workflow using the BalanceBot to characterize soft tissue balance, and the Apex Revision knee implant type
  Arms: Revision Total Knee Arthroplasty

SUMMARY:
This is a post-market multicentre study that has been implemented to confirm safety and performance of cemented CR/UC and PS Apex Knee implants in primary or revision Robotic Assisted Total Knee Arthroplasty up to 10-year follow up.

DETAILED DESCRIPTION:
This study has been implemented to confirm safety and performance of cemented CR/UC and PS Apex Knee implants in primary or revision RA-TKA up to 10-year follow up.

Prospective data will be collected for this Post Market Clinical Follow up (PMCF) study and the data will be fed into the Post-Market Surveillance (PMS) and Clinical Evaluation processes of the devices under assessment on annual basis and support presentations at orthopaedic congresses and/or peer-reviewed publication(s).

Participants will be selected for recruitment into the study from the general population of participants requiring a primary or revision knee-arthroplasty and considered suitable to receive the Apex Knee System.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be a candidate for a primary or revision total knee arthroplasty
2. Patient is able and willing to sign the informed consent and follow study procedures
3. Patient's joint must be anatomically and functionally suited to receive the selected implant and accommodate use of the robotic assistance

Exclusion Criteria:

1. Patient has a BMI >45.
2. Significant neurological or musculoskeletal disorders or disease that may interfere with total knee arthroplasty survival, adversely affect gait or weight bearing, (i.e. Paget's disease, Charcot's disease, muscular dystrophy, multiple sclerosis).
3. The presence of highly communicable disease or diseases that may limit follow-up (e.g. immuno-compromised conditions, hepatitis, active tuberculosis, HIV, etc.).
4. Presence of known active metastatic or neoplastic disease.
5. Cancer patients unless they have received curative treatment and have no evidence of recurrence for 5 years.
6. Patient has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease).
7. Patient has an active infection or joint sepsis.
8. Patient has muscular, neurological or vascular deficiencies which compromise the affected extremity (i.e., Parkinson's Disease, Multiple Sclerosis, and Charcot joints).
9. Patients with allergies or suspected sensitivity to any patient-contacting component of the implant to be used in the study Has known sensitivity to implants or the materials in the device including but not limited to: Ti, Al, V, Co, Cr, Mo, Ni and Si3N4.).
10. Patients who are currently on medical leave from their employment due to Worker's Compensation.
11. Patients who are at high risk for poor healing or confounding outcomes or at excessive risk for surgery (e.g., clinically significant/being actively treated for renal, hepatic, cardiac, hematologic, or neurologic disease or poorly controlled diabetes (HbA1c > 8 mg/dL) or previous history of joint infection).
12. Patients who are known drug or alcohol abusers or with psychological disorders as defined by DSM V that could affect follow-up care or treatment outcomes.
13. Patients who are currently involved in another clinical study with an investigational device.
14. Patients with current litigation pending related to medical treatment of any sort.
15. Patients, who, in the opinion of the investigator, will not be able to complete the study per the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 713 (Estimated)
Dates: Start 2017-11-09 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2040-04-01 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 Years
  Frequency of device and implant related adverse events and revision surgery to be recorded.

SECONDARY OUTCOMES:
Change in KOOS from baseline to 10 years after surgery | from enrolment to 10 years
  Evaluate impact of participants knee surgery, comparing post-operative Knee Injury and Osteoarthritis Outcome Score (KOOS) Scores and participants opinion about their knee
  KOOS ranges from 0 - 100, in which 100 is best.
Change in UCLA from baseline to 10 years after surgery | from enrolment to 10 years
  Evaluate impact of participants knee surgery, comparing post-operative Knee Injury and University of California Los Angeles (UCLA) activity Scale and measured the participants usual level of activity
  UCLA ranges from 0 - 10, in which the higher the score the greater the activity
Change in Promis-10 from baseline to 10 years after surgery | from enrolment to 10 years
  Evaluate impact of participants knee surgery, comparing post-operative Knee Injury and Patient-Reported Outcomes Measurement Information System (PROMIS) and measures the participants physical, mental, and social health.
  PROMIS-10 ranges from 1 - 67, in which 67 is best.

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Koenig, MD, Principal Investigator — NYU LANGONE-LONG ISLAND; Jeffrey H DeClaire, MD, Principal Investigator — DeClaire LaMacchia Orthopaedic Institute; Amber Randall, MD, Principal Investigator — Granite Orthopaedics; Corey Ponder, MD, Principal Investigator — Oklahoma Sports and Orthopedics Institute; John Keggi, MD, Principal Investigator — Orthopaedics New England; Jeffrey Lawrence, MD, Principal Investigator — Gundersen Lutheran Medical Foundation, Inc
Locations (6):
- United States (6):
  - Flagstaff Bone and Joint, Flagstaff, Arizona
  - Orthopaedics New England, Middlebury, Connecticut
  - DeClaire LaMacchia Orthopaedic Institute, Rochester, Michigan
  - Nyu Langone-Long Island, Garden City, New York
  - Oklahoma Sports and Orthopedics Institute, Oklahoma City, Oklahoma
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No